CLINICAL TRIAL: NCT00000464
Title: Cardiac Arrest in Seattle: Conventional Versus Amiodarone Drug Evaluation (CASCADE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: no record in DORA; R01HL031472 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Arrhythmia; Cardiovascular Diseases; Heart Arrest; Heart Diseases; Myocardial Infarction; Ventricular Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Arrest; Heart Diseases; Myocardial Infarction; Ventricular Fibrillation | interventions — Amiodarone; Imipramine; Mexiletine; Procainamide; Propafenone; Quinidine; Sotalol

INTERVENTIONS:
Drug: amiodarone
Drug: imipramine
Drug: mexiletine
Drug: procainamide
Drug: propafenone
Drug: quinidine
Drug: sotalol

SUMMARY:
To compare the efficacy of amiodarone to conventional anti-arrhythmic therapy in individuals who had survived one episode of out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
BACKGROUND:

Sudden cardiac death can usually be attributed to the occurrence of the cardiac arrhythmia, ventricular fibrillation. Although a significant proportion of patients experiencing sudden cardiac death may be successfully resuscitated without disabling sequelae, this event tends to recur. Recurrent sudden cardiac death is more common among patients demonstrating certain clinical characteristics such as: ventricular fibrillation occurring in a setting of a remote prior transmural infarction; the presence of abnormal left ventricular function; male gender; concurrent complex ventricular arrhythmias identified by electrocardiographic monitoring; extensive coronary artery disease; and the ability to induce ventricular arrhythmias following electrical stimulation.

Multiple therapeutic approaches are offered to patients surviving primary ventricular fibrillation. In those with evidence of myocardial ischemia, coronary revascularization procedures may be employed. Pharmacological therapy with anti-arrhythmic agents either alone or in combination with selection guided by the results of continuous electrocardiographic monitoring or electrophysiologic studies is often the initial step. For those patients refractory to medical therapy, ventricular resection or implantation of pacemakers has been employed.

Amiodarone, a unique antiarrhythmic agent with complex pharmacokinetics and substantial potential toxicity, has been utilized when other antiarrhythmic agents failed. The agent was released as an oral agent for the treatment of ventricular fibrillation in the United States by the FDA. Several investigations suggested that amiodarone was efficacious in the treatment of ventricular fibrillation when other available agents had failed.

DESIGN NARRATIVE:

Patients were stratified by presence or absence of coronary artery disease, left ventricular function, and presence or absence of drug failure prior to randomization. All patients underwent an evaluation of left ventricular ejection fraction, usually by radionuclide ventriculography, and baseline drug-free Holter recording or electrophysiologic study, or both. A total of 113 patients were randomized to amiodarone and 115 patients to conventional therapy with other antiarrhythmic agents which included procainamide, quinidine, disopyramide, tocainide, mexiletine, encainide, flecainide, propafenone, moricizine, or combination therapy in that order. Holter exams were given at one, three, six, twelve, twenty-four, and thirty-six months. Patients were followed for one to five years, with an average of three years overall. Primary endpoints for the study included in the term 'cardiac survival' were cardiac mortality, resuscitated cardiac arrest due to documented ventricular fibrillation, and complete syncope followed by a shock from an automated implanted defibrillator. These endpoints included sudden arrhythmic cardiac death, resuscitated out-of-hospital ventricular fibrillation, and nonarrhythmic cardiac death. A patient death due to amiodarone pulmonary toxicity was also considered a primary endpoint.

ELIGIBILITY:
Men and women with ventricular fibrillation who had survived an out-of-hospital cardiac arrest not associated with a Q-wave acute myocardial infarction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1987-04; Primary Completion 1992-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Greene — University of Washington

REFERENCES:
- [Background] Cardiac Arrest in Seattle: Conventional Versus Amiodarone Drug Evaluation (the CASCADE study). Am J Cardiol. 1991 Mar 15;67(7):578-84. doi: 10.1016/0002-9149(91)90895-r. PMID 2000790
- [Background] Greene HL. Sudden arrhythmic cardiac death--mechanisms, resuscitation and classification: the Seattle perspective. Am J Cardiol. 1990 Jan 16;65(4):4B-12B. doi: 10.1016/0002-9149(90)91285-e. PMID 2404396
- [Background] Poole JE, Mathisen TL, Kudenchuk PJ, McAnulty JH, Swerdlow CD, Bardy GH, Greene HL. Long-term outcome in patients who survive out of hospital ventricular fibrillation and undergo electrophysiologic studies: evaluation by electrophysiologic subgroups. J Am Coll Cardiol. 1990 Sep;16(3):657-65. doi: 10.1016/0735-1097(90)90357-u. PMID 2387939
- [Background] Dolack GL, Callahan DB, Bardy GH, Greene HL. Signal-averaged electrocardiographic late potentials in resuscitated survivors of out-of-hospital ventricular fibrillation. Am J Cardiol. 1990 May 1;65(16):1102-4. doi: 10.1016/0002-9149(90)90321-q. PMID 2330894
- [Background] Bardy GH, Allen MD, Mehra R, Johnson G, Feldman S, Greene HL, Ivey TD. Transvenous defibrillation in humans via the coronary sinus. Circulation. 1990 Apr;81(4):1252-9. doi: 10.1161/01.cir.81.4.1252. PMID 2317907
- [Background] Bardy GH, Troutman C, Johnson G, Mehra R, Poole JE, Dolack GL, Kudenchuk PJ, Gartman DM. Electrode system influence on biphasic waveform defibrillation efficacy in humans. Circulation. 1991 Aug;84(2):665-71. doi: 10.1161/01.cir.84.2.665. PMID 1860210
- [Background] Randomized antiarrhythmic drug therapy in survivors of cardiac arrest (the CASCADE Study). The CASCADE Investigators. Am J Cardiol. 1993 Aug 1;72(3):280-7. doi: 10.1016/0002-9149(93)90673-z. PMID 8342505
- [Background] Dolack GL. Clinical predictors of implantable cardioverter-defibrillator shocks (results of the CASCADE trial). Cardiac Arrest in Seattle, Conventional versus Amiodarone Drug Evaluation. Am J Cardiol. 1994 Feb 1;73(4):237-41. doi: 10.1016/0002-9149(94)90226-7. PMID 8296753
- [Background] Greene HL. The CASCADE Study: randomized antiarrhythmic drug therapy in survivors of cardiac arrest in Seattle. CASCADE Investigators. Am J Cardiol. 1993 Nov 26;72(16):70F-74F. doi: 10.1016/0002-9149(93)90966-g. PMID 8237833
- [Background] Maynard C. Rehospitalization in surviving patients of out-of-hospital ventricular fibrillation (the CASCADE Study). Cardiac Arrest in Seattle: Conventional Amiodarone Drug Evaluation. Am J Cardiol. 1993 Dec 1;72(17):1295-300. doi: 10.1016/0002-9149(93)90300-2. PMID 8256707